CLINICAL TRIAL: NCT07215455
Title: Efficacy And Safety of KSM66 Ashwagandha (Withania Somnifera) Standardized Root Extract (300 mg) on Weight and Stress Management in Overweight and Obese Adults: A Prospective, Randomized, Double-Blind Placebo- Controlled Study
Brief Title: Ashwagandha Extract for Weight and Stress Management in Overweight and Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SF Research Institute, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ixoreal-Weight-CT-03-23
Record Dates: First submitted 2025-10-02; First posted 2025-10-10 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Weight Management; Stress
MeSH Terms: interventions — Ashwagandha

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm 1: KSM-66 capsules containing Ashwagandha 300 mg standardized root extract. (Active Comparator): Ashwagandha 300 mg root extract in a dose of 300 mg capsules orally twice daily after breakfast and dinner with a glass of water or milk for 12 weeks.
  Interventions: Dietary Supplement: Ashwagandha 300 mg standardized root extract
- Treatment Arm 2: Identical placebo capsule. (Placebo Comparator): Identical Placebo in a dose of 300 mg capsules orally twice daily after breakfast and dinner with a glass of water or milk for 12 weeks.
  Interventions: Other: Identical placebo capsule.

INTERVENTIONS:
Dietary Supplement: Ashwagandha 300 mg standardized root extract — Participants in this group will receive KSM-66 Ashwagandha, a standardized root extract of Withania somnifera, 300 mg once daily in capsule form. KSM-66 is a high-concentration, full-spectrum extract of Ashwagandha root, designed to provide adaptogenic effects for stress reduction and support weight management. Participants will be instructed to take the capsule with water, preferably at the same time each day, for the duration of the 8-week study. Adherence will be monitored via pill counts and participant diaries.
  Arms: Treatment Arm 1: KSM-66 capsules containing Ashwagandha 300 mg standardized root extract.
Other: Identical placebo capsule. — Participants in this group will receive an identical placebo capsule that matches the appearance, size, color, and taste of the KSM-66 Ashwagandha capsule but contains inactive ingredients. The placebo is administered once daily for 8 weeks. Participants will be instructed to take the capsule with water, preferably at the same time each day. Adherence will be monitored via pill counts and participant diaries. The use of a placebo allows comparison with the Ashwagandha group to evaluate efficacy and safety outcomes while maintaining blinding for participants and study staff.
  Arms: Treatment Arm 2: Identical placebo capsule.

SUMMARY:
This study is designed to evaluate the effects of KSM-66 Ashwagandha root extract (300 mg daily) on weight management and stress reduction in overweight and obese adults. Ashwagandha (Withania somnifera) is a traditional herbal supplement that may help reduce stress and support overall health. In this randomized, double-blind, placebo-controlled trial, participants will receive either Ashwagandha extract or a placebo for the study duration. The main goal is to measure changes in body weight and stress levels. Other health outcomes, such as body mass index (BMI), waist circumference, and quality of life, will also be assessed. The study will help determine whether Ashwagandha is effective and safe for managing stress and supporting weight loss in adults with overweight or obesity.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled clinical study is being conducted to investigate the potential efficacy and safety of KSM-66 Ashwagandha® root extract (300 mg per capsule) in promoting weight management and reducing stress in adults classified as overweight or obese.

Participants will be randomly assigned to receive either KSM-66 Ashwagandha® capsules or matching placebo capsules for the study duration. Each participant will undergo baseline and follow-up assessments that include anthropometric measurements (body weight, BMI, and waist circumference), psychological evaluations (Perceived Stress Scale and related questionnaires), and laboratory investigations relevant to metabolic and stress-related health.

The study hypothesis is that daily supplementation with KSM-66 Ashwagandha® will lead to a statistically significant reduction in stress levels and body weight compared to placebo. The trial outcomes are expected to contribute to the growing body of evidence supporting the role of Ashwagandha as a safe and natural adaptogenic supplement for weight and stress management in adults.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult men and women participants ≥ 19 years and ≤65 years of age.
2. Willingness to follow the protocol requirements as evidenced by written informed consent.
3. Participants willing to give meaningful, written informed consent prior to participation in the trial, in accordance with regulatory requirements.
4. Participants who agree to take investigational product (i.e., Till Week 8).
5. Participants with Body mass index between 25 and 39.9 kg/m2

Exclusion Criteria:

1. History of Alcohol or smoking abuse.
2. History of hypersensitivity to Ashwagandha
3. Taking nutritional or energy supplements, medication, or steroids,
4. Any history of drug abuse
5. Having any clinical abnormalities
6. Simultaneously participating in any other clinical trial or participated in the past three months
7. Participants who use medication for blood pressure, use beta-blockers, inhaled any beta-agonists, use any hormonal contraceptives, having a history of corticosteroid use within three months, participants under psychotropic medication within last 8 weeks
8. Participants diagnosed with any heart disease, diabetes, stroke, neurological disorders or depression.
9. Have clinically significant acute unstable hepatic, renal, cardiovascular, or respiratory disease that will prevent participation in the study.
10. Patients with depressive episode, panic disorder, social phobia, obsessive-compulsory disorder, alcohol dependency; schizophrenia and mania.
11. Patients with post traumatic disorder.
12. Have an established practice of meditation (as meditating for at least 20 minutes, three or more times per week) for three or more months.
13. Pregnant and lactating women
14. Participation in other clinical trials during previous 3 months
15. Any clinical condition, according to the investigator which does not allow safe fulfilment of clinical trial protocol.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-06-17 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Mean change in body weight and BMI | aseline (Visit 1/Screening/Enrolment), Week 4 (Visit 2), Week 12 (Visit 3/End of Study)
  Change from baseline in body weight (kg) and body mass index (BMI, kg/m²) will be assessed in overweight and obese adult participants at Week 4 and Week 12. Measurements will be performed using standardized calibrated equipment under consistent conditions at each visit.

SECONDARY OUTCOMES:
Mean change in Perceived Stress Scale (PSS-10) score | Baseline, Week 4, Week 12
  Change from baseline in PSS-10 scores, measuring perceived stress levels in overweight and obese adult participants, at Week 4 and Week 12.
Mean change in SF-12 Health Survey score | Baseline, Week 4, Week 12
  Change from baseline in SF-12 scores, evaluating physical and mental health-related quality of life in overweight and obese adult participants, at Week 4 and Week 12.
Mean change in SSS (Stress Symptom Scale) score | Baseline, Week 4, Week 12
  Change from baseline in SSS scores, assessing self-reported stress symptoms in overweight and obese adult participants, at Week 4 and Week 12.
Mean change in Food Cravings Questionnaire-Trait (FCQ-T) score | Baseline, Week 4, Week 12
  Change from baseline in FCQ-T scores, evaluating trait-level food cravings in overweight and obese adult participants, at Week 4 and Week 12.
Mean change in Complete Blood Count (CBC) | Baseline, Week 4, Week 12
  Change from baseline in hematological parameters including hemoglobin (g/dL), total leukocyte count (cells/µL), and platelet count (cells/µL) measured by automated hematology analyzer.
Number and proportion of Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) | 12-week treatment period
  All TEAEs and TESAEs occurring during the 12-week intervention period will be recorded and summarized by number and proportion of participants affected, severity, and relationship to study intervention.
Mean change in Lipid Profile | Baseline, Week 4, Week 12
  Change from baseline in serum lipid parameters including total cholesterol (mg/dL), HDL cholesterol (mg/dL), LDL cholesterol (mg/dL), and triglycerides (mg/dL) measured by enzymatic colorimetric method.
Mean change in Liver Function Test (LFT) | Baseline, Week 4, Week 12
  Change from baseline in liver function parameters including serum alanine aminotransferase (ALT; U/L), aspartate aminotransferase (AST; U/L), alkaline phosphatase (ALP; U/L), and total bilirubin (mg/dL) measured using automated biochemistry analyzer.
Mean change in Renal Function Test (RFT) | Baseline, Week 4, Week 12
  Change from baseline in renal function parameters including serum creatinine (mg/dL) and blood urea nitrogen (BUN; mg/dL) measured using automated biochemistry analyzer.
Mean change in Thyroid Function Parameters | Baseline, Week 4, Week 12
  Change from baseline in serum Thyroxine (T4; µg/dL), Triiodothyronine (T3; ng/dL), and Thyroid-Stimulating Hormone (TSH; µIU/mL) measured by chemiluminescent immunoassay.
Mean change in Fasting Blood Sugar (FBS) | Baseline, Week 4, Week 12
  Change from baseline in fasting blood glucose level (mg/dL) measured by enzymatic glucose oxidase method.
Mean change in Glycated Hemoglobin (HbA1c) | Baseline, Week 4, Week 12
  Change from baseline in HbA1c (%) measured by high-performance liquid chromatography (HPLC).

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Research Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No